CLINICAL TRIAL: NCT05200481
Title: A Phase II Randomized, Open-Labelled, Multicenter Study of Safety & Efficacy of Combination Brigatinib and Carboplatin-Pemetrexed Therapy or Brigatinib Monotherapy as First-Line Treatment in Advanced ALK-Positive Non-Small Cell Lung Cancer
Brief Title: Study of Safety and Efficacy of Brigatinib Plus Chemotherapy or Brigatinib Only in Advanced ALK-Positive Lung Cancer (MASTERPROTOCOL ALK)
Acronym: MP-ALK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-2101
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer; ALK Gene Mutation
Keywords: IFCT; NCSLC; brigatinib; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib; Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Interventional, phase II, randomized, open-labelled, non-comparative multicenter study with two parallel arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brigatinib monotherapy Arm A (Other): Brigatinib 180mg QD (1 x 180mg tablet) until progression
  Interventions: Drug: Brigatinib 180 MG
- Brigatinib Carboplatin-Pemetrexed combination therapy Arm B (Experimental): Brigatinib 180mg QD (1 x 180mg tablet) until progression + Carboplatin AUC of 5 mg/mL/min IV infusion every 3 weeks for 4 infusions + pemetrexed 500 mg/m² IV infusion every 3 weeks for 4 infusions
  Interventions: Drug: Brigatinib 180 MG; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Brigatinib 180 MG — Patients will receive brigatinib orally at a dose of 90 mg QD for a 7 days lead-in period followed by 180 mg QD continuously, with or without food, in 28-day cycles until progression. Dose reductions are possible.
  Other Names: ALUNBRIG
Drug: Carboplatin — Patients will receive pemetrexed 500 mg/m² followed by carboplatin to target AUC of 5 mg/mL/min both on Day 1 as IV infusion every 3 weeks for 4 infusions. The first infusion of carboplatin and pemetrexed will be administrated at day 8 of brigatinib treatment, at time of dose escalation from 90 mg QD to 180mg QD continuously.
  Arms: Brigatinib Carboplatin-Pemetrexed combination therapy Arm B
Drug: Pemetrexed — Patients will receive pemetrexed 500 mg/m² followed by carboplatin to target AUC of 5 mg/mL/min both on Day 1 as IV infusion every 3 weeks for 4 infusions. The first infusion of carboplatin and pemetrexed will be administrated at day 8 of brigatinib treatment, at time of dose escalation from 90 mg QD to 180mg QD continuously.
  Arms: Brigatinib Carboplatin-Pemetrexed combination therapy Arm B

SUMMARY:
This is a phase II randomized, open-labelled, non-comparative multicenter study in which ALK+ NSCLC patients who are naïve of treatment for advanced disease will be randomized to receive brigatinib monotherapy (Arm A) or brigatinib and carboplatin-pemetrexed therapy (Arm B). An estimated 110 patients (55 in Arm A, 55 in Arm B) will be enrolled at approximately 30 centers. A safety phase will evaluate the safety of brigatinib with carboplatin and pemetrexed treatment combination (Arm B). The first twenty-six patients enrolled in Arm B will represent the population of the safety phase. Patients will be treated until they experience progressive disease, intolerable toxicity, or another discontinuation criterion is met. Continuation of brigatinib beyond progression is permitted, at the investigator's discretion, if there is evidence of continued clinical benefit. The null hypothesis is progression free survival at 12 months ≤ 69% for Arm B, which is considered not sufficiently clinically meaningful to warrant further study. The alternative hypothesis is that 86% or more of patients in Arm B would achieve progression free survival at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care. Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
2. Patients diagnosed with histologically or cytologically confirmed locally advanced not eligible to a local treatment or metastatic NSCLC (Stage IIIB, IIIC or IV accordingly to 8th classification TNM, UICC 2015).
3. Patients are eligible for trial entry on the basis of locally determined ALK testing. ALK Immunohistochemistry (IHC) assay (3+ only), DNA-based or RNA-based next generation sequencing (NGS) assay, nCounter Nanostring assay or ALK FISH performed locally are accepted ALK testing assays. If ALK rearrangement diagnostic is performed using IHC and the result is + or 2+, a confirmation with a second method performed locally (DNA-based or RNA-based NGS assay, nCounter Nanostring assay or ALK FISH performed) is required.
4. All Patients must have at least one measurable target lesion according to RECIST v1.1 per investigator assessment. The radiological assessment has to be done within the timelines indicated.
5. Patients with asymptomatic and neurologically stable CNS metastases (including patients controlled with less than 10mg/day of methylprednisolone within the last week prior to study entry) will be eligible.
6. Tumor Sample Requirement: sufficient tumor tissue for central analysis should be available (tumor block or a minimum of 10 unstained slides of 4 µm of analyzable tissue).
7. Age ≥18 years.
8. Life expectancy of at least 12 weeks, in the opinion of the Investigator.
9. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
10. Adequate Bone Marrow Function, including: Absolute Neutrophil Count (ANC) ≥1.5 x 109/L; Platelets ≥100 x 109/L; Hemoglobin ≥9 g/dL.
11. Adequate Pancreatic Function, including: Serum lipase ≤3.0 ULN.
12. Adequate Renal Function, including: Estimated creatinine clearance ≥45 mL/min as calculated using the standard method of the institution.
13. Adequate Liver Function, including: Total serum bilirubin ≤1.5 x ULN (<3.0 × ULN for patients with Gilbert syndrome); Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x ULN; ≤5.0 x ULN if there is liver metastases involvement.
14. Participants must have recovered from toxicities related to prior anticancer therapy to CTCAE Grade ≤ 1.
15. Participants must have recovered from effects of any major surgery, or significant traumatic injury, at least 35 days before the first dose of treatment.
16. Have normal QT interval on screening ECG evaluation, defined as QT interval corrected (QTc) of ≤450 milliseconds (msec) in males or ≤470 msec in females.
17. Female patients who: are postmenopausal for at least 1 year before the screening visit, OR are surgically sterile, OR if they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, one of them being nonhormonal, from the time of signing the informed consent through 6 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
18. Male patients, even if surgically sterilized (i.e., status post-vasectomy), who: agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
19. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedure.
20. Participant has national health insurance coverage.

Exclusion Criteria:

1. Previously received an investigational antineoplastic agent for NSCLC.
2. Previously received any prior TKI, including ALK-targeted TKIs.
3. Known molecular co-alteration i.e. activating EGFR/BRAF/KRAS/MET mutation and ROS1/RET/NTRK fusion.
4. Previously received neo-adjuvant or adjuvant systemic chemotherapy or consolidation immunotherapy if completion of (neo) adjuvant/consolidation therapy occurred <12 months prior to randomization.
5. Patients who have leptomeningeal disease (LM) or carcinomatous meningitis (CM) according to MRI data and/or in case of documented cerebral spinal fluid (CSF) positive cytology.
6. Spinal cord compression.
7. Patients with symptomatic or neurologically instable CNS metastases.
8. Major surgery within 30 days of study entry. Minor surgical procedures (e.g., port insertion, mediastinoscopy, surgical procedure for re-sampling) are not excluded, but sufficient time at investigator discretion should have passed for wound healing.
9. Radiation therapy within 2 weeks of study entry. Stereotactic or small field brain irradiation must have completed at least 2 weeks prior to study entry. Whole brain radiation must have completed at least 4 weeks prior to study entry.
10. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
11. Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to: a) myocardial infarction within 6 months prior to the first dose of study drug; b) unstable angina within 6 months prior to the first dose of study drug; c) congestive heart failure within 6 months prior to the first dose of study drug; d) any history of ventricular arrhythmia; e) history of clinically significant atrial arrhythmia or clinically significant bradyarrhythmia as determined by the treating physician; f) cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose of study drug.
12. Have uncontrolled hypertension. Patients with hypertension should be under treatment on study entry to control blood pressure.
13. History of grade 3 or 4 of interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, pulmonary fibrosis and radiation pneumonitis.
14. Presence of interstitial fibrosis of any grade at baseline.
15. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
16. Evidence of active malignancy (other than current NSCLC, non-melanoma skin cancer, in situ cervical cancer, papillary thyroid cancer, DCIS of the breast or localized and presumed cured prostate cancer) within the last 3 years.
17. Active inflammatory gastrointestinal disease, malabsorption syndrome, chronic diarrhea, symptomatic diverticular disease or previous gastric resection or lap band.
18. Current use or anticipated need for food or drugs prohibited.
19. Patients presenting with abnormal Left Ventricular Ejection Fraction (LVEF) by echocardiogram or Multi-Gated Acquisition Scan (MUGA) according to institutional lower limits.
20. Have a known or suspected hypersensitivity to brigatinib, carboplatin or pemetrexed or their excipients.
21. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
22. Received systemic treatment with strong cytochrome p-450 (cyp)3a inhibitors, strong cyp3a inducers, or moderate cyp3a inducers within 14 days before enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 12 months, investigator assessment | 12 months
  Time from enrollment to first observation of progression (RECIST1.1) or date of death (from any cause), determined by investigator assessment.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) at 12 months, independent review | 12 months
  Time from enrollment to first observation of progression (RECIST1.1) or date of death (from any cause), determined by independent review.
Overall Response Rate (ORR) | At progression, after an average of 2 years
  Proportion of patients who have achieved a best overall response of complete response or partial response (RECIST1.1), determined by investigator assessment and by independent review.
Incidence, nature, and severity of adverse events | From time of informed consent through treatment period and up to 30 days post last dose of study treatment (average of 2 years)
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0).
Impact of ALK fusion detection in ctDNA on 12-months progression free survival | 12 months
  Proportion of patients who achieved progression free survival (RECIST1.1) with ALK fusion detection in ctDNA baseline liquid biopsy, determined by investigator assessment and by independent review.
Impact of ALK fusion detection in ctDNA on overall response rate | At progression, after an average of 2 years
  Proportion of patients who have achieved a best overall response of complete response or partial response (RECIST1.1) with ALK fusion detection in ctDNA baseline liquid biopsy, determined by investigator assessment and by independent review.
Intracranial overall response rate | At progression, after an average of 2 years
  Proportion of patients who have achieved a best overall response of complete response or partial response of the baseline measurable and non-measurable CNS disease (RECIST1.1 + RANO), determined by investigator assessment and by independent review.
Intracranial progression free survival at 12 months | 12 months
  Proportion of patients achieving an objective response (CR or PR) of the baseline measurable and non-measurable CNS disease according to RECIST 1.1 and Revised Assessment in Neuro Oncology (RANO) criteria, determined by investigator assessment and by independent review.
Time until definitive health related quality of life score deterioration | From enrollment to score deterioration, a period of up to 2 years
  The European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30/QLQ-LC13 questionnaire will be used to determine time until definitive HRQoL score deterioration.
Duration of response (DOR) | At progression, after an average of 2 years.
  Time from the date of first documented response (CR or PR) to the earliest date of disease progression (RECIST1.1), determined by investigator assessment and by independent review.
Disease control rate (DCR) | At progression, after an average of 2 years.
  Proportion of patients who have achieved a confirmed best overall response of CR, PR or SD (RECIST v1.1), determined by investigator assessment and by independent review.
Overall survival (OS) | At death or lost to follow up, up to 5 years after randomisation.
  Time between the date of randomization and death or last date of follow-up.
Duration of intracranial response (CNS DOR) | At progression, after an average of 2 years.
  Time from the first occurrence of an objective response (CR or PR) of the baseline measurable and non-measurable CNS disease for at least 12 weeks, according to RECIST 1.1. and Revised Assessment in Neuro Oncology (RANO) criteria, determined by investigator assessment and independent review.
Intracranial disease control rate (CNS DCR) | At progression, after an average of 2 years.
  Proportion of patients achieving a response (CR, PR or SD) of the baseline measurable and non-measurable CNS disease according to RECIST 1.1 and Revised Assessment in Neuro Oncology (RANO) criteria, determined by investigator assessment and independent review.

CONTACTS AND LOCATIONS:
Overall Officials: Michael DURUISSEAUX, Dr, Principal Investigator — Hospices Civils de Lyon - Hôpital Louis Pradel; Aurélie SWALDUZ, Dr, Principal Investigator — Centre Leon Berard
Locations (29):
- France (29):
  - CHU d'Angers, Angers
  - CHU Besançon - Hôpital J. MINJOZ, Besançon
  - Hôpital APHP Ambroise Paré, Boulogne
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron
  - CHU Côte de Nacre, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Georges-François Leclerc, Dijon
  - Chu Grenoble, Grenoble
  - Hôpital Calmette, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Nord, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier, Mulhouse
  - Hôpital Cochin, Paris
  - Hôpital BICHAT, Paris
  - Hôpital TENON, Paris
  - Hôpital Haut-Lévèque, Pessac
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain
  - Centre Hospitalier, Saint-Quentin
  - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - HIA Sainte-Anne, Toulon
  - Hôpital Larrey (CHU), Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Centre Hospitalier de Villefranche-sur-Saône, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/